CLINICAL TRIAL: NCT03186287
Title: Effectiveness of Eccentric and Concentric Strength Training in Patients With Subacromial Impingement Syndrome: A Randomized Controlled Trial
Brief Title: Effectiveness of Eccentric and Concentric Strength Training in Patients With Subacromial Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Damla Karabay, MSc, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2837-GOA
Record Dates: First submitted 2017-06-09; First posted 2017-06-14 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Subacromial Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Eccentric training group (Experimental): The participants in this group will actively perform eccentric phase of resistive shoulder exercises. Additionally they will receive standard physiotherapy.
  Interventions: Other: Eccentric training; Other: Standard physiotherapy
- Concentric training group (Experimental): The participants in this group will actively perform concentric phase of resistive shoulder exercises. Additionally they will receive standard physiotherapy.
  Interventions: Other: Concentric training; Other: Standard physiotherapy
- Control group (Active Comparator): The participants in this group will receive only standard physiotherapy.
  Interventions: Other: Standard physiotherapy

INTERVENTIONS:
Other: Eccentric training — Eccentric phase of resistive shoulder exercises will be performed three sets of 15 repetitions once a day for 12 weeks using therabands. Participants will be supervised by the physiotherapist 3 days a week for the first 6 weeks, 2 days a week for the next 3 weeks and 1 day a week for the last 3 weeks.
  Arms: Eccentric training group
Other: Concentric training — Concentric phase of resistive shoulder exercises will be performed three sets of 15 repetitions once a day for 12 weeks using therabands. Participants will be supervised by the physiotherapist 3 days a week for the first 6 weeks, 2 days a week for the next 3 weeks and 1 day a week for the last 3 weeks.
  Arms: Concentric training group
Other: Standard physiotherapy — The participants will receive standard physiotherapy. The standard physiotherapy exercises will be supervised by the physiotherapist, same as intervention exercises.

SUMMARY:
The purpose of this study is to investigate and compare the effects of eccentric and concentric strength training on pain, strength, joint position sense and function in patients with subacromial impingement syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of subacromial impingement syndrome
* Complaints associated with subacromial impingement syndrome for at least 3 months
* No extra pain with 90 degree abduction-90 degree external rotation position of the shoulder
* Ability to complete the entire study procedure

Exclusion Criteria:

* Severe pain; shoulder pain is > 7/10
* History of upper extremity fracture
* History of shoulder, cervical and thoracic surgery
* Having shoulder instability or frozen shoulder diagnosis
* History of shoulder injuries, trauma and / or shoulder symptoms requiring treatment during the last 1 year (except than subacromial impingement syndrome)
* Full-thickness rotator cuff tear
* Systemic musculoskeletal disease
* Neck and shoulder pain with cervical spine movement
* Chest deformity or scoliosis diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Shoulder Function | Baseline, 12 weeks and 24 weeks
  Change of Constant Murley Score

SECONDARY OUTCOMES:
Pain intensity | Baseline, 12 weeks and 24 weeks
  Change of visual analog scale score in activity and rest
Upper extremity function | Baseline, 12 weeks and 24 weeks
  Change of disabilities of the arm, shoulder, and hand (DASH) score
Isometric strength | Baseline, 12 weeks and 24 weeks
  Change of shoulder abduction and external rotation isometric strength (in kg, with hand held dynamometer)
Eccentric strength | Baseline, 12 weeks and 24 weeks
  Change of shoulder abduction and external rotation eccentric strength (in kg, with hand held dynamometer)
Joint position sense | Baseline, 12 weeks and 24 weeks
  Change of shoulder joint repositioning angle errors (with bubble inclinometer)

CONTACTS AND LOCATIONS:
Overall Officials: Damla KARABAY, MSc, Principal Investigator — Izmir Katip Celebi University; Sevgi Sevi YESILYAPRAK, PhD, Study Director — Dokuz Eylul University; Mehmet ERDURAN, MD, Study Director — Dokuz Eylul University; Cem OZCAN, MD, Study Director — Izmır Katip Celebi University Atatürk Training and Research Hospital
Locations (1):
- Dokuz Eylul University, School of Physical Therapy and Rehabilitation, Izmir, Balçova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No